CLINICAL TRIAL: NCT05430633
Title: Laparoscopic Versus Open Appendectomy in Pregnancy. 10 Year Results of Estonian Population.
Brief Title: Laparoscopic Versus Open Appendectomy in Pregnancy
Status: Completed | Type: Observational
Sponsor: North Estonia Medical Centre (Other)
Responsible Party: Principal Investigator, Edgar Lipping, Principal investigator, general surgeon, MD, North Estonia Medical Centre
Other Study IDs: 345T-2
Record Dates: First submitted 2022-06-12; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Appendicitis; Pregnancy Loss; Pregnancy Preterm
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant patients who underwent laparoscopic appendectomy: Pregnant patients who underwent laparoscopic appendectomy
  Interventions: Procedure: Appendectomy
- Pregnant patients who underwent open appendectomy: Pregnant patients who underwent open appendectomy
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy — Appendectomy - laparoscopic or open

SUMMARY:
The aim of this retrospective trial is to compare surgical and pregnancy outcomes of pregnant patients who underwent laparoscopic or open appendectomy for acute appendicitis.

DETAILED DESCRIPTION:
The aim of this retrospective trial is to compare surgical and pregnancy outcomes of pregnant patients who underwent laparoscopic or open appendectomy for acute appendicitis.

Patients' medical records from 2010-2020 were extracted using billing information of the national health insurance fund of Estonia and ICD-10 codes (pregnancy, appendicitis).

Collected data was stored on RedCap electronic database and analyzed with R Studio.

Two group of patients were compared: pregnant patients who had laparoscopic appendectomy and pregnant patients who had open appendectomy.

ELIGIBILITY:
Inclusion Criteria:

Women with confirmed pregnancy who underwent appendectomy for acute appendicitis.

Exclusion Criteria:

Women who were not pregnant when having an appendectomy

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Study population consists of pregnant women who were pregnant during appendectomy confirmed either before or after the surgical procedure. The population was derived from the billing information from years 2010-2020 of the national health insurance fund of Estonia.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Obstetrical outcomes | Pregnancy loss within 9 months from appendectomy
  Pregnancy loss (fetal demise) - rate of cessation of pregnancy before scheduled delivery

SECONDARY OUTCOMES:
Surgical outcomes | 30 days after appendectomy
  Surgical complications - rate of infectious complications within 30 days after appendectomy

CONTACTS AND LOCATIONS:
Locations (1):
- North Estonia Medical Centre, Tallinn, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee SH, Lee JY, Choi YY, Lee JG. Laparoscopic appendectomy versus open appendectomy for suspected appendicitis during pregnancy: a systematic review and updated meta-analysis. BMC Surg. 2019 Apr 25;19(1):41. doi: 10.1186/s12893-019-0505-9. PMID 31023289
- [Background] Prodromidou A, Machairas N, Kostakis ID, Molmenti E, Spartalis E, Kakkos A, Lainas GT, Sotiropoulos GC. Outcomes after open and laparoscopic appendectomy during pregnancy: A meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2018 Jun;225:40-50. doi: 10.1016/j.ejogrb.2018.04.010. Epub 2018 Apr 9. PMID 29656140
- [Background] Zeng Q, Aierken A, Gu SS, Yao G, Apaer S, Anweier N, Wu J, Zhao JM, Li T, Tuxun T. Laparoscopic Versus Open Appendectomy for Appendicitis in Pregnancy: Systematic Review and Meta-Analysis. Surg Laparosc Endosc Percutan Tech. 2021 May 3;31(5):637-644. doi: 10.1097/SLE.0000000000000943. PMID 33935257